CLINICAL TRIAL: NCT07027397
Title: One Year of Velocity-based Resistance Training in Older People Living in Nursing Homes: Effects on Skeletal Muscle Mass, Muscle Function, and Physical and Cognitive Function
Brief Title: One Year of Velocity-based Resistance Training in Older People Living in Nursing Homes
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Castilla-La Mancha (Other)
Responsible Party: Principal Investigator, Julián Alcázar Caminero, PhD, Associate Professor, University of Castilla-La Mancha
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 710P
Record Dates: First submitted 2025-05-27; First posted 2025-06-18 (Actual); Last update posted 2025-06-18 (Actual); Status verified 2025-05

CONDITIONS: Aging; Muscle Mass and Strength; Muscle Power; Frailty Syndrome; Cognitive Function
MeSH Terms: conditions — Frailty | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Exercise Group (Experimental): a 2-day-a-week resistance training (RT) routine using the velocity-based method in the leg press exercise at 60% of the theoretical maximal isometric strength
  Interventions: Other: Exercise

INTERVENTIONS:
Other: Exercise — All participants will conduct a 2-day-a-week resistance training (RT) routine using the velocity-based method in the leg press exercise for one year. A tailored and constant intensity will be performed at 60% of the theoretical maximal isometric strength (F0) during the training intervention. Participants will conduct 3-4 sets, individualizing the repetitions numbers until they reach a velocity loss of 10-20%. A rest of 2 minutes was imposed between sets. A standardized warm-up will preced all RT session as follows: 4 minutes walking at usual gait speed and 6 minutes performing dynamic balance exercises.

SUMMARY:
This study is an exercise intervention assessing the efficacy of a velocity-based resistance training (VBRT) in institutionalized older adults.

The aim of this study is to assess the effects of one year of velocity-based resistance training on skeletal muscle mass, muscle function, and physical and cognitive function in older adults living in nursing homes.

DETAILED DESCRIPTION:
Evidence supports the fact that resistance exercise training is effective in improving old adult's health and palliate age-related disorders. New approaches in resistance training are emerging to maximize monitoring control, providing more tailored and potentially more effective exercise interventions. Among them, the velocity-based resistance training (VBRT) is being established in healthy populations or populations with pathologies. However, the effects of long-term VBRT in institutionalized older adults are still unknown.

Thus, the aim of this study is to assess the effects of one year of velocity-based resistance training on skeletal muscle mass, muscle function, and physical and cognitive function in older adults living in nursing homes.

ELIGIBILITY:
Inclusion Criteria:

* Older people living permanently in nursing home.
* Age ≥ 65 years old.
* Are able to walk with/without assistance.
* Have ability to communicate with the research team.

Exclusion Criteria:

* Terminal illness.
* Any illness not controled (cardiac, pulmonary, etc).
* If there is a risk of bone fracture according to medical staff.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2024-09-30 (Actual); Primary Completion 2024-12-05 (Actual); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Change in muscle power | T0 (baseline); T1 (post 6 weeks); T2 (post 12 weeks); T3 (post 23 weeks) and T4 (post 39 weeks).
  Muscle power assessed in leg press machine and sit to stand test.
Changes in neuromuscular performance of lower-body | T0 (baseline); T1 (post 6 weeks); T2 (post 12 weeks); T3 (post 23 weeks) and T4 (post 39 weeks).
  Change in the force-velocity relationship in leg press exercise.

SECONDARY OUTCOMES:
Change in physical function based on the Short Physical Performance Battery score | T0 (baseline); T1 (post 6 weeks); T2 (post 12 weeks); T3 (post 23 weeks) and T4 (post 39 weeks).
  The Short Physical Performance Battery score ranges from 0 to 12 points. Higher scores indicate better physical function, while lower scores reflect poorer physical function.
Change in frailty (score) using Fried's Frailty Criteria and Frailty Trait Scale - Short Form | T0 (baseline); T1 (post 6 weeks); T2 (post 12 weeks); T3 (post 23 weeks) and T4 (post 39 weeks).
  Fried's frailty phenotype based on five criteria (habitual gait speed, handgrip strength , involuntary weight loss, exhaustion and low physical activity). The score ranges from 0 to 5, where each criterion met counts as one point. A score of 0 indicates best status, while a score of 5 indicates worst status.
  Frailty Trait Scale - Short Form evaluates 5 domains, including body mass index, physical activity, static balance, habitual gait speed and handgrip strength. The score ranges from 0 to 50, where each criterion met counts as one point. A score of 0 indicates best status, while a score of 50 indicates worst status.
Change in muscle mass using ultrasonography. | T0 (baseline); T1 (post 6 weeks); T2 (post 12 weeks); T3 (post 23 weeks) and T4 (post 39 weeks).
  Muscle Cross-sectional area quadriceps femoris were assessed using ultrasonography.
Change in disability using Barthel and Lawton scales | T0 (baseline); T1 (post 6 weeks); T2 (post 12 weeks); T3 (post 23 weeks) and T4 (post 39 weeks).
  The Lawton scale assesses the ability to use the telephone, shopping, cooking, household duties, laundry, use of transportation, responsibility for their medication and handling of economic matters. Each item is assigned a numerical value (1 = independent, 0 = dependent), therefore, the maximum dependence would be marked by obtaining 0 points (worst) and total independence by obtaining 8 points (best).
  The Barthel index is a 10-item questionnaire that provides information about the autonomy to cook food, wash, dress, groom, perform bowel movements and urination, go to the toilet, move from the bed to the chair, walk and climb stair.The total score ranges from 0 to 100, with higher scores indicating greater independence (best), and lower scores indicating higher levels of dependence in basic daily activities (worst).
Change in cognitive function using Mini-Mental State Examination | T0 (baseline); T1 (post 6 weeks); T2 (post 12 weeks); T3 (post 23 weeks) and T4 (post 39 weeks).
  Mini-Mental State Examination score ranges from 0 to 30 points. A higher score indicates better cognitive function, while a lower score reflects greater cognitive impairment.
Change in handgrip strength | T0 (baseline); T1 (post 6 weeks); T2 (post 12 weeks); T3 (post 23 weeks) and T4 (post 39 weeks).
  Change in maximum voluntary isometric handgrip strength, measured using a digital dynamometer.

CONTACTS AND LOCATIONS:
Overall Officials: Julian Alcazar, PhD, Principal Investigator — University of Castilla-La Mancha
Locations (1):
- University of Castilla-La Mancha, Toledo, Toledo, Spain